CLINICAL TRIAL: NCT02886117
Title: Creation and Evaluation of a Auto-administered Questionnaire by Screening of Disorder of the Haemostasis in Preoperative
Brief Title: Auto-administered Questionnaire by Screening of Disorder of the Haemostasis in Preoperative
Acronym: HEMOSTASE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TROUBLE HEMOSTASE (RB 14.121)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Preoperative Assessment of Hemostasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to determine the capacity of a questionnaire to predict a normal balance sheet of haemostasis.

DETAILED DESCRIPTION:
Recent recommendations formalized by experts of the French society of anaesthesiology on systematic pre-interventional examinations recommend assessing the risk of bleeding from personal and family history of bleeding diathesis and after physical examination . They recommend not to prescribe a systematic hemostasis laboratory tests in patients with a history and physical examination do not suspect a disorder of hemostasis.

However, there is currently no validated questionnaire in the general population to assess the preoperative bleeding risk allowing a reliable assessment of the personal and family bleeding diathesis.

The establishment of a structured questionnaire, the patient could filled before surgery consultation to guide the possible prescription of a balance sheet, could meet the new recommendations.

It seems therefore important to establish this type of questionnaire in order to optimize the operation of the structure, and to limit the requirements of routine hemostasis balance sheets. To do this, the investigator wants to carry out a preliminary study to ensure the interest of the established questionnaire.

The questionnaire assessed in this study is drawn from existing specialized questionnaires, the description of hemostasis disorders described factor for deficits from the doctor in charge of hemophilia expertise center and expertise of a psychologist, to refine best.

ELIGIBILITY:
Inclusion Criteria:

* All adults addressed in programmed anesthesia consultation, regardless of whether surgery and consultation site

Exclusion Criteria:

* Patients minors
* Physical or mental disability in Patient to agree and complete the questionnaire
* Major patients undergoing a protective measure
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population coming in programmed anesthesia consultation
Sampling Method: Non-Probability Sample
Enrollment: 2511 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
hemostasis tests (normal or abnormal) | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Yves Ozier, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France